CLINICAL TRIAL: NCT07121608
Title: Exploring Dental Anxiety in Patients With Special Needs: A Randomised Cross-over Study of I-MDAS and Malay Version of MDAS
Brief Title: Exploring Dental Anxiety in Special Needs Patients: A Comparison of I-MDAS and Malay MDAS
Acronym: MDAS
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Aisyah Ahmad Fisal, Dental Lecturer (Special Care Dentistry), University of Malaya
Other Study IDs: DF CD2308/0019/2447 (P); UMG045E-2024 (Other Grant/Funding Number: Dental Postgraduate Research Grant)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Dental Anxiety
Keywords: Randomised cross-over; Patients with special needs; Dental anxiety; Modified Dental Anxiety Scale; Acceptability; Special Care Dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (M-MDAS → I-MDAS): Participants in this group will first complete the Malay Modified Dental Anxiety Scale (M-MDAS) in the initial session. After a one-week washout period, they will then complete the Inclusive Modified Dental Anxiety Scale (I-MDAS), which includes video, narration, and subtitles for improved accessibility.
- Group B (I-MDAS → M-MDAS): articipants in this group will begin by completing the Inclusive Modified Dental Anxiety Scale (I-MDAS) in the first session. Following a one-week washout period, they will complete the Malay Modified Dental Anxiety Scale (M-MDAS) in the second session.

SUMMARY:
This study aims to better understand and improve how dental anxiety is measured in patients with special needs (PSN) who visit the Special Care Dentistry (SCD) Clinic at Universiti Malaya (UM). Researchers want to find out:

Whether there is a difference in anxiety scores when using two versions of a dental anxiety questionnaire - the Inclusive Modified Dental Anxiety Scale (I-MDAS) and the Malay Modified Dental Anxiety Scale (M-MDAS).

Which version PSN prefer or find easier to use. What factors may cause higher dental anxiety in these patients. What factors are linked to more severe levels of dental anxiety.

Participants in this study will be randomly assigned to one of two groups. Each group will try out two different versions of a dental anxiety questionnaire - the written Malay Modified Dental Anxiety Scale (M-MDAS) and the Inclusive Modified Dental Anxiety Scale (I-MDAS), which includes video and narration.

First, participants will fill out a short questionnaire about their background, such as age, gender, education, medical history, and dental experiences.

Then, depending on their group, they will complete either the M-MDAS or the I-MDAS first.

After a one-week break (called a "washout period"), they will complete the other version of the questionnaire.

This allows researchers to compare both tools fairly and see which one is more effective and preferred by patients with special needs.

DETAILED DESCRIPTION:
This study is designed to improve how dental anxiety is measured in patients with special needs (PSN) who receive care at the Special Care Dentistry (SCD) Clinic at Universiti Malaya (UM). Dental anxiety can make it harder for patients to visit the dentist, especially those with disabilities or complex medical conditions. To support better care, researchers want to understand which assessment method works best for this group.

The study focuses on two versions of a dental anxiety questionnaire:

I-MDAS (Inclusive Modified Dental Anxiety Scale) - a video-based tool with narration and subtitles to make it more accessible.

M-MDAS (Malay Modified Dental Anxiety Scale) - a standard written version in the Malay language.

The study will explore:

Whether there are differences in anxiety scores between I-MDAS and M-MDAS. Which version is easier for PSN to understand and complete. What personal, medical, or dental history factors are linked to higher or more severe dental anxiety.

What Will Participants Do?

Participants will first complete a pre-questionnaire about their background, including age, gender, education, type of special care needs, medical history, when they last saw a dentist, and whether they've had any unpleasant dental experiences.

Participants will then be randomly assigned to one of two groups:

Group A will complete the M-MDAS first, followed by I-MDAS. Group B will complete the I-MDAS first, followed by M-MDAS. There will be a one-week washout period between the two sessions to reduce any influence from the first questionnaire on the second.

After completing both tools, participants will also be asked which version they found easier or more comfortable to use.

By comparing the two tools and collecting feedback from PSN, the researchers aim to recommend a more inclusive and effective way to measure dental anxiety in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. New and existing patients attending SCD clinic at Faculty of Dentistry, Universiti Malaya for elective dental treatment
3. Literate and able to understand the Malay language
4. Frankl behavioural rating scale of score 3 and 4

Exclusion Criteria:

1. Patients who require other urgent dental treatments
2. Severe or complex learning or ID
3. Frankl behavioural rating scale of score 1 and 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with special needs attending Special Care Dentistry Clinic at Faculty of Dentistry, Universiti Malaya
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Agreement Between I-MDAS and M-MDAS in Measuring Dental Anxiety | Within 2 weeks of enrolment (completion of both I-MDAS and M-MDAS with 1-week washout period)
  This outcome measures the level of agreement between the Inclusive Modified Dental Anxiety Scale (I-MDAS) and the Malay Modified Dental Anxiety Scale (M-MDAS) in assessing dental anxiety among patients with special needs (PSN). Agreement will be evaluated using statistical methods such as the intraclass correlation coefficient (ICC), Bland-Altman plot, and paired comparisons of total scores from both tools.

SECONDARY OUTCOMES:
Acceptability of I-MDAS Compared to M-MDAS | Immediately after completion of both anxiety scales (within 2 weeks of enrolment)
  Acceptability will be measured using a structured questionnaire consisting of five Likert-scale items (1 = strongly disagree to 5 = strongly agree) that assess participants' agreement with statements about their experience using the Malay Modified Dental Anxiety Scale (M-MDAS) and the Inclusive Modified Dental Anxiety Scale (I-MDAS). Items assess ease of understanding, usability, comfort, satisfaction, and future preference. The total acceptability score for each version will be calculated and compared between tools. Preference for I-MDAS over M-MDAS will also be captured through a forced-choice item.
Factors Associated With Severity of Dental Anxiety (I-MDAS Scores) | At baseline (upon initial assessment during first visit)
  This outcome investigates demographic, medical, and dental-related factors linked to the severity of dental anxiety, as measured by the I-MDAS total score. Statistical analyses such as multiple linear regression and group comparisons (e.g., ANOVA or Kruskal-Wallis) will be used to identify associations.
  The I-MDAS is scored on a scale from 5 to 25, with higher scores indicating greater levels of dental anxiety (i.e., a worse outcome).
Factors Associated With Presence of Dental Anxiety (I-MDAS) | At baseline (upon initial assessment during first visit)
  This outcome identifies sociodemographic and clinical characteristics that are associated with the presence of dental anxiety (based on a defined cut-off score on the I-MDAS). Chi-square tests, Fisher's exact tests, and logistic regression will be used to explore associations between participant factors and anxiety status.
  The I-MDAS is scored on a scale from 5 to 25, with higher scores indicating greater levels of dental anxiety (i.e., a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Aisyah Ahmad Fisal, BDS, MSCD RCSEd, D.Ch.Dent SCD, Principal Investigator — Dental Lecturer (Special Care Dentistry)
Locations (1):
- Special Care Dentistry Clinic, Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share individual participant data (IPD). The dataset will not be made publicly available due to concerns about participant privacy and data sensitivity in a special needs population.